CLINICAL TRIAL: NCT00735943
Title: Macugen Observational Study
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5751031
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2011-08-16 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Vascular Endothelial Growth Factor; Macular Degeneration
Keywords: Pegaptanib; macular degeneration; vascular endothelial growth factor
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The objective of this observational study is to evaluate the effectiveness and safety of Macugen for treatment of wet age-related macular degeneration (AMD) in Indian patients.Prospective, Observational, Non-interventional Study. The period of observation for the study will be 1 year

DETAILED DESCRIPTION:
To be eligible for enrollment in this study, patients must receive the first injection of Macugen intravitreal in at least one eye for treatment of wet age-related macular degeneration (AMD). The decision to prescribe Macugen will necessarily precede and will be independent of the decision to enroll patient into the study.

If both eyes of a patient receive injection Macugen, only one eye will be included in the study. If both eyes receive first injection Macugen after initiation of the study, only the first treated eye will be included in the analysis. If one eye has already received Macugen when the study starts and the second eye receives injection after the study initiation, the second eye will be included in the analysis.

The study was prematurely discontinued due to delay in meeting pre-defined protocol recruitment milestones on August 30, 2010. There were no safety concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for enrollment in this study, patients must receive the first injection of Macugen intravitreal in at least one eye for treatment of wet age-related macular degeneration (AMD).

Exclusion Criteria:

* Active or suspected ocular or periocular infection.
* Known hypersensitivity to pegaptanib sodium or any other excipient in this product.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be eligible for enrollment in this study, patients must receive the first injection of Macugen intravitreal in at least one eye for treatment of wet age-related macular degeneration (AMD).
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- India (5):
  - Pfizer Investigational Site, Navrangpura, Ahemdabad, Gujarat
  - Pfizer Investigational Site, Gurgaon, Haryana
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Jaipur, Rajasthan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751031&StudyName=Macugen%20Observational%20Study%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegaptanib: Macugen 0.3 mg (pegaptanib sodium) administered once every 6 weeks by intravitreal injection into the study eye.
Period: Overall Study
Arm/Group | Pegaptanib
Started | 22
Completed | 20
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pegaptanib
Number analyzed (Participants) | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 70.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Showing Stabilization, Improvement or Deterioration of Visual Acuity (VA)
Description: VA was measured using ETDRS (Early Treatment Diabetic Retinopathy Study) chart at 4 meter distance, at 1 meter distance (if participant's VA was poor) or verifying if the participant was able only to count fingers, to perceive hand motion or light. VA was assessed as the number of ETDRS letters correctly read. VA statuses were defined as: Stabilization: loss of less than 15 letters in the best corrected VA (BCVA); Improvement: gain of more than or equal to 15 letters in the BCVA; Deterioration: loss of more than or equal to 15 letters in the BCVA.
Time Frame: Baseline through 12 months or last follow-up visit before study termination
Population: Full Analysis Set (FAS) included all participants who received at least 1 injection of the study treatment in the study eye during the study. Missing values were imputed by Last Observation Carried Forward (LOCF) technique.
Measure: Number; unit: percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 22
percentage of participants
  Improvement | 18.2
  Stabilization | 54.5
  Deterioration | 18.2

2. Primary Outcome: Average Number of Injections to Achieve Stabilization of VA
Description: Stabilization of VA was defined as loss of less than 15 letters in the BCVA. For each participant, number of injections before reaching the first "stabilization in VA" (considered as an event) was counted. For participant having no event, the time to the number of injections to reach an event was unobserved at the number of injections before the last follow up.
Time Frame: 12 months or last follow-up visit before study termination
Population: FAS included all participants who received at least 1 injection of the study treatment in the study eye during the study. Missing values were imputed by LOCF technique. Analysis was conducted for those participants who received at least 1 injection of the study treatment in the study eye and achieved stabilization at the last follow-up.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Pegaptanib
Number analyzed (Participants) | 12
injections | 2.25 (1.14)

3. Primary Outcome: Median Number of Injections to Achieve Stabilization of VA
Description: Stabilization of VA was defined as loss of less than 15 letters in the BCVA. Median number of injections to achieve stabilization of VA was estimated via the Kaplan Meier method. For each participant, number of injections before reaching the first "stabilization in VA" (considered as an event) was counted. For participant having no event, the time to the number of injections to reach an event was unobserved at the number of injections before the last follow up.
Time Frame: 12 months or last follow-up visit before study termination
Population: as for outcome 2
Measure: Median (Full Range); unit: injections
Arm/Group | Pegaptanib
Number analyzed (Participants) | 12
injections | 2.00 [1.00 to 4.00]

4. Secondary Outcome: Percentage of Participants Receiving Macugen Monotherapy Versus Those Receiving a Combination Therapy
Description: Macugen monotherapy: referred to participants receiving Macugen in the study eye during the study that is (i.e.) participants without any concomitant drug treatment or nondrug treatment for the study eye during the study. Combination therapy: referred to participants receiving combination therapy in the study eye (during the study) i.e. participants with any concomitant drug treatment or nondrug treatment for the study eye during the study.
Time Frame: 12 months or last follow-up visit before study termination
Population: FAS included all participants who received at least 1 injection of the study treatment in the study eye during the study. Missing values were imputed by LOCF analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 22
Percentage of participants
  Macugen monotherapy | 100
  Combination therapy | 0

5. Secondary Outcome: Percentage of Participants Showing Improvement in Optical Coherence Tomography (OCT) Parameters
Description: OCT, a noninvasive, noncontact, transpupillary imaging technology, was utilized to image retinal structures in vivo with a resolution of 10 to 17 microns. The anatomic layers within the retina, retinal thickness could be measured. Improvement in OCT parameters was defined as a reduction of more than or equal to 100 microns in the central macular thickness (Center subfield).
Time Frame: 12 months or last follow-up visit before study termination
Population: FAS included all participants who received at least 1 injection of the study treatment in the study eye during the study. Missing values were imputed by LOCF technique.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 22
Percentage of participants
  Improvement | 13.6
  No improvement | 54.5
  Lost to follow up | 27.3
  No 'center subfield' value | 4.5

6. Secondary Outcome: Percentage of Participants Showing Improvement in Fundus Fluorescein Angiography (FFA) Parameters
Description: A fluorescein angiogram provides information about the condition of the retina. Improvement in FFA parameters was defined as absence of progression of the lesion or decrease in the size of the lesion and absence of new lesions on FFA i.e. change in lesion size from baseline must be less than or equal to 0 disc area(DA) and no new lesions.
Time Frame: 12 months or last follow-up visit before study termination
Population: Due to small sample size, the analysis was not conducted.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants With Early Lesions Showing Stabilization and Improvement of VA
Description: Early lesions were defined by any 2 of the following criteria: occult lesion diagnosed on FFA; baseline VA of more than or equal to 54 ETDRS letters; lesion size of less than 2DA on FFA. Stabilization of VA was defined as loss of less than 15 letters in the BCVA. Improvement in the VA was defined as gain of more than or equal to 15 letters in the BCVA.
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

8. Secondary Outcome: Average Number of Injections to Achieve Stabilization of VA in Participants With Early Lesions
Description: as for outcome 2
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Number; unit: injections
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

9. Secondary Outcome: Median Number of Injections to Achieve Stabilization of VA in Participants With Early Lesions
Description: Stabilization of VA was defined as loss of less than 15 letters in the BCVA. Median number of injections to achieve stabilization of VA in participants with early lesions was estimated via the Kaplan Meier method. For each participant, number of injections before reaching the first "stabilization in VA" (considered as an event) was counted. For participant having no event, the time to the number of injections to reach an event was unobserved at the number of injections before the last follow up.
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Median (Full Range); unit: injections
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With Occult or Minimally Classic and Classic Lesions Showing Stabilization and Improvement in VA
Description: FFA was utilized to characterize the lesions as follows: Classic lesion: more than 50% of the lesion had a well-demarcated area of hyperfluorescence; minimally classic lesion: less than or equal to 50% of lesion had well-demarcated area of hyperfluorescence; occult lesion: lesion with no well demarcated borders. VA statuses were defined as: stabilization: loss of less than 15 letters in the BCVA; improvement: gain of more than or equal to 15 letters in the BCVA.
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants Who Were Treatment Naive When Started on Macugen Versus Those Previously Treated by Any Other Therapy Except Macugen
Description: Participants were considered treatment naive when started on Macugen and without any previous drug or non drug treatment administered to the study eye. Participants were considered previously treated by any other therapy if received any other drug or non drug treatment to the study eye except Macugen.
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

12. Secondary Outcome: Percentage of Participants Showing Stabilization or Improvement in VA in the Subgroup Previously Treated by Other Therapy
Description: VA was measured using ETDRS chart at 4 meter distance, at 1 meter distance (if patient's VA was poor) or verifying if the patient was able only to count fingers, to perceive hand motion or light. VA was measured as the number of ETDRS letters correctly read. VA statuses were defined as: stabilization: loss of less than 15 letters in the BCVA; improvement: gain of more than 15 letters in the BCVA.
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of Participants Showing Improvement in OCT in the Subgroup Previously Treated by Other Therapy
Description: OCT, a noninvasive, noncontact, transpupillary imaging technology, was utilized to image retinal structures in vivo with a resolution of 10 to 17 microns. The anatomic layers within the retina, retinal thickness could be measured. Improvement in OCT parameters was defined as a reduction of more than or equal to 100 microns in the central macular thickness (Center subfield). Improvement in OCT parameters was measured based on this single parameter.
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants Showing Improvement in OCT in the Subgroup Which Were Not Treatment Naive
Description: as for outcome 13
Time Frame: 12 months or last follow-up visit before study termination
Population: Subgroup analysis was not performed as the study was terminated due to slow rate of recruitment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pegaptanib
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegaptanib (N=22)
Retinal haemorrhage (Eye disorders) | 1 (2)
Visual acuity reduced (Eye disorders) | 1 (2)
Subretinal fibrosis (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Outcome measures were not designated as primary or secondary measures as this study was an observational non-interventional study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.